CLINICAL TRIAL: NCT02108717
Title: The Feasibility Study for Remote CT Reading for Suspected Acute Appendicitis Using iPhone With Remote Control System in Realtime Under the Ambient Bright.
Brief Title: The Feasibility Study for Real-time Remote CT Reading for Suspected Acute Appendicitis Using iPhone
Acronym: Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Changsun Kim, Clinical assistant professor, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-02
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Telemedicine
Keywords: Telemedicine; appendicitis; remote consultation
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): The raters in this group one firstly reviewed the CT scans numbered from one to 60 using LCD monitor and after mandatory rests of 20 minutes, reviewed the remaining CT examinations numbered from 61 to 120 using iPhone with TeamViewer at their first visit.
  They visited twice with an interval of four weeks and reviewed the CT scans using revered devices at each session.
  Interventions: Device: Remote CT reading using the iPhone; Device: CT reading using LCD monitor
- Group II (Experimental): The raters in this group II firstly reviewed the CT scans numbered from one to 60 using iPhone with TeamViewer and 61 to 120 with the LCD monitor.
  They visited twice with an interval of four weeks and reviewed the CT scans using revered devices at each session.
  Interventions: Device: Remote CT reading using the iPhone; Device: CT reading using LCD monitor

INTERVENTIONS:
Device: Remote CT reading using the iPhone
  Other Names: Smartphone (A1530, iPhone 5S, USA)
Device: CT reading using LCD monitor
  Other Names: LCD monitor (MX210, EIZO, Japan)

SUMMARY:
1. Purpose

   - The investigators aim to evaluate the feasibility of iPhone based remote control system as a real-time remote CT reading tool for suspected appendicitis under 3G network and the suboptimal illumination.
2. Methods

   * A total of 120 abdominal CT examinations; sixty had no findings of appendicitis, while the other sixty showed signs of acute appendicitis, were selected. The 16 raters reviewed these images using an LCD monitor of the PACS workstation and also an iPhone which was connected to the PACS workstation via remote control system, grading the probability of presence of acute appendicitis on each examination by a five Likert scale.
   * The investigators will compare the diagnostic performance between two devices.

DETAILED DESCRIPTION:
The 16 raters were randomly divided into two groups

* The raters in group one reviewed the CT examinations numbered from one to 60 using LCD monitor and reviewed the remaining CT examinations numbered from 61 to 120 using iPhone with TeamViewer at their first visit
* The other group firstly reviewed the CT scans numbered from one to 60 using iPhone with TeamViewer and 61 to 120 with the LCD monitor.
* They visited twice with an interval of four weeks and reviewed the CT scans using revered devices at each session.
* The raters were instructed to rate the likelihood of the presence or absence of appendicitis in each case using a five-Likert scale (1 = obvious no appendicitis, 2 = unlikely appendicitis, 3 = unsure, 4 = likely appendicitis, 5 = obvious appendicitis).

ELIGIBILITY:
Inclusion Criteria:

* Board certified emergency physicians with a clinical experience of 5 years and over.

Exclusion Criteria:

* Corrected eyesight < 20/30
* Color weakness or blindness

Ages: 33 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance between iPhone and LCD monitor | within one day
  * Dorfman-Berbaum-Metz method with RSCORE and semi-parametric estimation of ROC indices by using the DMB-MRMC software (version 2.3, available at http://perception.radiology.uiowa.edu)
  * 95% confidence interval
  * The reviewers and cases are taken as random factors
Diagnostic accuracy between the iPhone and the LCD monitor | within one day
  ◆ Sensitivity, specificity
  * gold standard: The pathology report and the results of clinical follow up
  * grade 1, 2 and 3 = negative appendicitis findings
  * grade 4 and 5 = positive appendicitis findings
  * McNemar's test to compare the sensitivity and specificity between the iPhad and the LCD monitor

CONTACTS AND LOCATIONS:
Overall Officials: Bo Seung Kang, MD, Study Director — Hanyang University Guri Hospital
Locations (1):
- Hanyang university guri hospital, Department of emergency medicine, Guri-si, GyeongGido, South Korea

REFERENCES:
- [Background] Choi HJ, Lee JH, Kang BS. Remote CT reading using an ultramobile PC and web-based remote viewing over a wireless network. J Telemed Telecare. 2012 Jan;18(1):26-31. doi: 10.1258/jtt.2011.110412. Epub 2011 Nov 8. PMID 22067287
- [Background] Choudhri AF, Carr TM 3rd, Ho CP, Stone JR, Gay SB, Lambert DL. Handheld device review of abdominal CT for the evaluation of acute appendicitis. J Digit Imaging. 2012 Aug;25(4):492-6. doi: 10.1007/s10278-011-9431-9. PMID 22146833
- [Background] Park JB, Choi HJ, Lee JH, Kang BS. An assessment of the iPad 2 as a CT teleradiology tool using brain CT with subtle intracranial hemorrhage under conventional illumination. J Digit Imaging. 2013 Aug;26(4):683-90. doi: 10.1007/s10278-013-9580-0. PMID 23404630
- [Derived] Kim C, Kang B, Choi HJ, Park JB. A Feasibility Study of Real-Time Remote CT Reading for Suspected Acute Appendicitis Using an iPhone. J Digit Imaging. 2015 Aug;28(4):399-406. doi: 10.1007/s10278-015-9775-7. PMID 25700617
- See also: Displaymate: Flagship Smartphone Display Technology Shoot-Out — http://www.displaymate.com/Smartphone_ShootOut_2.htm
- See also: Hayes JC. Monitor's megapixels do not affect image interpretation — http://www.diagnosticimaging.com/conference-reports/scar2005/article/113619/1198917